CLINICAL TRIAL: NCT06331156
Title: A Phase III, Open-label, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of Inactivated Poliovirus Vaccine (IPV) When Co-administered With Porcine Circovirus (PCV)-Free Liquid Formulation of an Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Chinese Infants
Brief Title: A Study on the Immune Response and Safety of Inactivated Poliovirus Vaccine (IPV) When Co-administered With Human Rotavirus (HRV) Porcine Circovirus (PCV)-Free Vaccine in Healthy Chinese Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 218485; 2022-000708-36 (EudraCT Number)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteritis
Keywords: Human rotavirus (HRV); Rotarix Porcine circovirus (PCV)-free liquid; Inactivated poliovirus vaccine (IPV); Healthy Chinese infants; Immunogenicity; Safety
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-administration Group (Experimental): Participants received 2 doses of PCV-free liquid formulation of GSK's oral live attenuated HRV vaccine co-administered with the first 2 doses of IPV vaccine at Month 0.5 and Month 1.5, followed by the third dose of IPV vaccine administered at Month 2.5.
  Interventions: Combination Product: HRV PCV-free; Combination Product: IPV
- Staggered Group (Active Comparator): Participants received 2 doses of Porcine circovirus (PCV)-free liquid formulation of GSK's oral live attenuated human rotavirus (HRV) vaccine at Day 1 and Month 1, and 3 doses of Inactivated poliovirus vaccine (IPV) vaccine administered at Month 0.5, Month 1.5, and Month 2.5.
  Interventions: Combination Product: HRV PCV-free; Combination Product: IPV

INTERVENTIONS:
Combination Product: HRV PCV-free — 2 doses of HRV PCV-free vaccine are administered orally at Month 0.5 and Month 1.5 (Co-administration Group) and at Day 1 and Month 1 (Staggered Group), according to the immunization schedule for HRV vaccine licensed outside of China. PCV-free implies no detection of PCV-1 and PCV-2 according to the limit of detection of the tests used.
  Other Names: Rotarix PCV-free
Combination Product: IPV — 3 doses of IPV vaccine are administered intramuscularly at Month 0.5, Month 1.5 and Month 2.5 (Co-administration Group and Staggered Group), according to the recommended schedule for vaccination against poliovirus in China.
  Other Names: Beijing Biological Products Institute Co.,Ltd.'s Inactivated Poliomyelitis Vaccine Made From Sabin Strains (Vero Cells)

SUMMARY:
The purpose of this study is to evaluate the immune response and safety of the inactivated poliovirus (IPV) vaccine when co-administered with the human rotavirus (HRV) porcine circovirus (PCV)-free vaccine in healthy Chinese infants 6-10 weeks of age at the time of study enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/Legally Acceptable Representative(s) [LAR(s)], who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female of Chinese origin, between and including, 6 and 10 weeks (42-76 days) of age at the time of study enrolment.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* History of severe combined immunodeficiency.
* History of seizures or progressive neurological disease.
* Family history of congenital or hereditary immunodeficiency.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception (IS).
* History of IS.
* Major congenital defects, or serious chronic illness as assessed by the investigator.
* Any contraindications to IPV.
* Previous confirmed occurrence of rotavirus gastroenteritis (RVGE).
* History of poliomyelitis.
* Participants with confirmed or suspected Coronavirus Disease 2019 (COVID-19).

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days before the first dose of study interventions (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of study interventions administration*, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study and other licensed routine childhood vaccinations.

  *In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
* Administration of long-acting immune-modifying drugs from birth or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives from birth or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone >=0.5 milligram/kilogram (kg)/day, or equivalent. Inhaled, intra-articular and topical steroids are allowed.
* Previous vaccination against RV.
* Previous vaccination against poliomyelitis.

Prior/Concurrent clinical study experience

- Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.

Other exclusions

- Child in care.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - GSK Investigational Site, Mianyang
  - GSK Investigational Site, Neijiang
  - GSK Investigational Site, Wenshan
  - GSK Investigational Site, Yuechi-Guang'an

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in China.
Pre-assignment Details: A total of 400 participants were included in Enrolled set, out of which only 392 were included in Exposed set and started the study.
Period: Overall Study
Arm/Group | Staggered Group | Co-administration Group
Started | 199 | 193
Completed | 186 | 189
Not Completed | 13 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Migrated / Moved from the study area | 4 | 3
Not completed — Other | 7 | 0
Not completed — Adverse event requiring expedited reporting | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Staggered Group | Co-administration Group | Total
Number analyzed (Participants) | 199 | 193 | 392
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.1 (1.2) | 8.2 (1.3) | 8.1 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 92 | 188
  Male | 103 | 101 | 204
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 199 | 193 | 392

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion for Anti-poliovirus Types 1, 2 and 3 Neutralizing Antibody (Ab)
Description: Seroconversion for anti-poliovirus types 1, 2 and 3 neutralizing Ab is defined as: - Ab titer greater than or equal to (>=) 1:8 at 1 month after the 3 dose primary vaccination schedule of IPV in participants with Ab titer lower than (<) 1:8 at pre-vaccination, >= 4-fold increase in Ab titer at 1 month after the 3 dose primary vaccination schedule of IPV in participants with Ab titer >= 1:8 at pre-vaccination.
Time Frame: At Month 3.5 (1 month post-Dose 3 of IPV)
Population: Analysis was performed on the per protocol set (PPS) for IPV, comprising participants who adhered to their assigned intervention schedule without conditions affecting immunogenicity or using prohibited treatments. For anti-poliovirus types 1, 2, and 3 at 1 month post-Dose 3, participants must have pre- and post-vaccination immunogenicity data for at least one antigen and adhered to the interval between Dose 3 and blood sample at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 125 | 143
Percentage of participants
  anti-poliovirus serotype1 | 99.2 [95.6 to 100] | 99.3 [96.2 to 100]
  anti-poliovirus serotype2 | 100 [97.1 to 100] | 99.3 [96.2 to 100]
  anti-poliovirus serotype3 | 100 [97.1 to 100] | 100 [97.5 to 100]
Statistical Analysis 1: Comparison: Staggered Group vs Co-administration Group; To demonstrate the immunological non-inferiority of IPV when co-administered with HRV PCV-free compared with IPV administered alone in terms of seroconversion rates 1-month post-Dose 3 of IPV (Month 3.5); Test type: Non-Inferiority — Non-inferiority (NI) was to be demonstrated if the lower limit (LL) of the 2-sided 95% confidence interval (CI) for the group difference (Co-administration group minus Staggered group) in seroconversion rate is greater than or equal to (>=) -10% for the anti-poliovirus type 1 antibodies; Difference in seroconversion rate = 0.10, 95% CI 2-sided [-3.14 to 3.76] — The asymptotic standardized 95% CI for the difference in seroconversion rate for IPV at month 3.5 between Co-administration group minus staggered group is computed using the method of Miettinen and Nurminen
Statistical Analysis 2: Comparison: Staggered Group vs Co-administration Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — NI was to be demonstrated if the LL of the 2-sided 95% CI for the group difference (Co-administration group minus Staggered group) in seroconversion rate is >= -10% for the anti-poliovirus type 2 antibodies; Difference in seroconversion rate = -0.70, 95% CI 2-sided [-3.86 to 2.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Staggered Group vs Co-administration Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — NI was to be demonstrated if the LL of the 2-sided 95% CI for the group difference (Co-administration group minus Staggered group) in seroconversion rate is >= -10% for the anti-poliovirus type 3 antibodies; Difference in seroconversion rate = 0.00, 95% CI 2-sided [-2.63 to 2.99] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Anti-poliovirus Types 1, 2 and 3 Neutralizing Ab
Time Frame: At Month 3.5 (1 month post-Dose 3 of IPV)
Population: Analysis was performed on the PPS for IPV. Only participants with data available at the specified timepoints were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 125 | 143
Titers
  anti-poliovirus serotype1 | 1369.71 [1140.65 to 1644.78] | 1374.44 [1148.21 to 1645.25]
  anti-poliovirus serotype2 | 194.95 [168.13 to 226.06] | 190.44 [164.90 to 219.94]
  anti-poliovirus serotype3 | 451.36 [389.37 to 523.23] | 450.15 [395.92 to 511.79]

3. Secondary Outcome: Percentage of Participants With Anti-poliovirus Types 1, 2 and 3 Neutralizing Ab Titers >=1:8 and >=1:64
Time Frame: At Month 3.5 (1 month post-Dose 3 of IPV)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 125 | 143
Percentage of participants
  anti-poliovirus serotype1, >=1:8 | 100 [97.1 to 100] | 100 [97.5 to 100]
  anti-poliovirus serotype1, >=1:64 | 100 [97.1 to 100] | 100 [97.5 to 100]
  anti-poliovirus serotype2, >=1:8 | 100 [97.1 to 100] | 100 [97.5 to 100]
  anti-poliovirus serotype2, >=1:64 | 91.2 [84.8 to 95.5] | 91.6 [85.8 to 95.6]
  anti-poliovirus serotype3, >=1:8 | 100 [97.1 to 100] | 100 [97.5 to 100]
  anti-poliovirus serotype3, >=1:64 | 98.4 [94.3 to 99.8] | 99.3 [96.2 to 100]

4. Secondary Outcome: Percentage of Participants With Seroconversion for Anti-rotavirus (RV) Immunoglobulin A (IgA) Ab
Description: Seroconversion for anti-RV IgA Ab is defined as: anti-RV IgA Ab concentration >= 20 unit per milliliter (U/mL) at 1 month post-Dose 2 of HRV PCV-free vaccine, in participants who were initially seronegative (i.e., with anti-RV IgA Ab concentration < 20 U/mL prior to the first dose of HRV PCV-free vaccine).
Time Frame: At 1 month post-Dose 2 of HRV PCV-free vaccine (Month 2 for Staggered Group and Month 2.5 for Co-administration Group)
Population: Analysis was performed on the PPS for RV, comprising participants who adhered to their assigned intervention schedule without conditions affecting immunogenicity or using prohibited treatments. For anti-RV IgA analyses at 1 month post Dose 2 of HRV PCV-free, participants should have pre- and post-vaccination immunogenicity results and should have complied with the interval between HRV Dose 2 and the post HRV PCV-free Dose 2 blood sample at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 130 | 146
Percentage of participants | 78.5 [70.4 to 85.2] | 90.4 [84.4 to 94.7]

5. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-RV IgA Ab
Time Frame: At 1 month post-Dose 2 of HRV PCV-free vaccine (Month 2 for Staggered Group and Month 2.5 for Co-administration Group)
Population: Analysis was performed on the PPS for RV. Only participants with data available at the specified timepoints were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 130 | 146
U/mL | 160.59 [114.49 to 225.25] | 222.15 [165.98 to 297.34]

6. Secondary Outcome: Percentage of Participants With Anti-RV IgA Ab Concentrations >= 90 U/mL
Time Frame: At 1 month post-Dose 2 of HRV PCV-free vaccine (Month 2 for Staggered Group and Month 2.5 for Co-administration Group)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 130 | 146
Percentage of participants | 63.8 [55.0 to 72.1] | 68.5 [60.3 to 75.9]

7. Secondary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: Solicited systemic events include cough/runny nose, diarrhoea, fever (pyrexia), irritability/fussiness, loss of appetite and vomiting. Fever is defined as body temperature >= 37.5 degrees Celsius (°C) and the preferred location for measuring temperature is the axilla. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Within 14 days after Dose 1 & 2: HRV PCV-free vaccine administered at Day 1 & Month 1 (Staggered group) and at Month 0.5 & Month 1.5 (Co-administration group); IPV administered at Month 0.5 & Month 1.5 (Staggered and Co-administration group)
Population: Analysis was performed on the Exposed set, which includes all participants who received at least one dose of any of the 2 study interventions and for whom solicited systemic events data were available after the corresponding vaccination for the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 197 | 193
Participants
  Cough/Runny Nose, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Cough/Runny Nose, post vaccination at Day 1 | 21 |
  Cough/Runny Nose, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Cough/Runny Nose, post vaccination at Month 0.5 | 28 | 27
  Cough/Runny Nose, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Cough/Runny Nose, post vaccination at Month 1 | 27 |
  Cough/Runny Nose, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Cough/Runny Nose, post vaccination at Month 1.5 | 23 | 22
  Diarrhoea, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Diarrhoea, post vaccination at Day 1 | 8 |
  Diarrhoea, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Diarrhoea, post vaccination at Month 0.5 | 10 | 9
  Diarrhoea, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Diarrhoea, post vaccination at Month 1 | 11 |
  Diarrhoea, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Diarrhoea, post vaccination at Month 1.5 | 7 | 12
  Fever, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Fever, post vaccination at Day 1 | 15 |
  Fever, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Fever, post vaccination at Month 0.5 | 46 | 23
  Fever, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Fever, post vaccination at Month 1 | 33 |
  Fever, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Fever, post vaccination at Month 1.5 | 25 | 21
  Irritability/Fussiness, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Irritability/Fussiness, post vaccination at Day 1 | 15 |
  Irritability/Fussiness, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Irritability/Fussiness, post vaccination at Month 0.5 | 11 | 19
  Irritability/Fussiness, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Irritability/Fussiness, post vaccination at Month 1 | 6 |
  Irritability/Fussiness, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Irritability/Fussiness, post vaccination at Month 1.5 | 6 | 7
  Loss of appetite, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Loss of appetite, post vaccination at Day 1 | 14 |
  Loss of appetite, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Loss of appetite, post vaccination at Month 0.5 | 10 | 20
  Loss of appetite, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Loss of appetite, post vaccination at Month 1 | 5 |
  Loss of appetite, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Loss of appetite, post vaccination at Month 1.5 | 5 | 4
  Vomiting, post vaccination at Day 1: number analyzed (Participants) | 197 | 0
  Vomiting, post vaccination at Day 1 | 12 |
  Vomiting, post vaccination at Month 0.5: number analyzed (Participants) | 192 | 193
  Vomiting, post vaccination at Month 0.5 | 6 | 18
  Vomiting, post vaccination at Month 1: number analyzed (Participants) | 191 | 0
  Vomiting, post vaccination at Month 1 | 6 |
  Vomiting, post vaccination at Month 1.5: number analyzed (Participants) | 189 | 191
  Vomiting, post vaccination at Month 1.5 | 1 | 7

8. Secondary Outcome: Number of Participants Reporting Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs include any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Within 31 days after each dose of HRV PCV-free vaccine (administered at Day 1 and Month 1 for Staggered Group and at Month 0.5 and Month 1.5 for Co-administration group)
Population: Analysis was performed on the Exposed set, which includes all participants who received at least one dose of any of the 2 study interventions and for whom unsolicited AEs data were available after the corresponding vaccination for the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 199 | 193
Participants
  HRV PCV-free: post-Dose 1 | 38 | 45
  HRV PCV-free: post-Dose 2: number analyzed (Participants) | 192 | 191
  HRV PCV-free: post-Dose 2 | 39 | 34

9. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or in other situations that are considered serious per medical or scientific judgment. Any = occurrence the event regardless of intensity grade or relation to the study vaccination.
Time Frame: From the first dose of the study intervention (Day 1 for Staggered group and Month 0.5 for Co-administration group) up to study end (Month 3.5)
Population: Analysis was performed on the Exposed set, which includes all participants who received at least one dose of any of the 2 study interventions and for whom SAE data were available after the corresponding vaccinations for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Staggered Group | Co-administration Group
Number analyzed (Participants) | 199 | 193
Participants | 30 | 30

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 14 days after Dose 1 & 2: HRV PCV-free vaccine administered at Day 1 & Month 1 (Staggered group) and at Month 0.5 & Month 1.5 (Co-administration group); IPV administered at Month 0.5 & Month 1.5 (Staggered and Co-administration group), Unsolicited AEs: Within 31 days after each dose of HRV PCV-free vaccine. All-cause mortality and SAEs were collected throughout the study period (From Day 1 to Month 3.5).
Description: SAEs, solicited AEs and unsolicited AEs were reported for the Exposed set.
Arm/Group | Staggered Group | Co-administration Group
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/193
Serious Adverse Events (participants affected / at risk) | 30/199 | 30/193
Other Adverse Events (participants affected / at risk) | 141/199 | 129/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Staggered Group (N=199) | Co-administration Group (N=193)
Pneumonia (Infections and infestations) | 17 (17) | 16 (17)
Febrile infection (Infections and infestations) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 3 (3) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 2 (2) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Secondary thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Staggered Group (N=199) | Co-administration Group (N=193)
Respiratory tract infection (Infections and infestations) | 66 (98) | 40 (49)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 9 (9)
Pharyngitis (Infections and infestations) | 6 (6) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 32 (36) | 25 (27)
Vomiting (Gastrointestinal disorders) | 18 (25) | 22 (25)
Constipation (Gastrointestinal disorders) | 6 (7) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 70 (78) | 50 (51)
Decreased appetite (Metabolism and nutrition disorders) | 28 (33) | 22 (26)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 30 (37) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 3 (3)
Myocardial injury (Cardiac disorders) | 2 (2) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT06331156/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT06331156/SAP_001.pdf